CLINICAL TRIAL: NCT07325019
Title: THE EFFECTS OF AEROBİC EXERCİSE ON NEUROVASCULAR UNİT AND CLİNİCAL PROGRESSİON MARKERS İN INDİVİDUALS WİTH MULTİPLE SCLEROSİS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Elif Asan, Advanced Physiotherapist, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024313
Record Dates: First submitted 2025-12-02; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Aerobic Exercise; Neurovascular Unit; Multiple Sclerosis; Biomarker; Clinical Progression
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Each patient was recommended a conventional exercise programme tailored to their needs. These included exercises aimed at strengthening the lower extremities and torso, exercises targeting patients' balance and walking problems (progressing from hard to soft surfaces, from eyes open to eyes closed, and from a wide support base to a narrow support base), walking training exercises (ceremonial walking, walking with reduced support area, sideways walking exercises), and exercises targeting coordination problems (Frenkel coordination exercises from sitting and supine positions, depending on the patient's condition).
- aerobic exercise (Active Comparator): The aerobic exercise programme was implemented over a total of 8 weeks, with two sessions per week, using a treadmill under the supervision of a specialist physiotherapist. Patients' functional capacities were determined by estimating VO2 peak using walking distance, heart rate, and blood pressure measured at 6 DYT. During the aerobic exercise programme, patients' heart rates and oxygen saturation levels were monitored using a pulse oximeter, and care was taken to ensure that the Borg Scale value perceived by patients was between 11 and 14. After the aerobic exercise programme ended, heart rate, blood pressure, and Borg Scale were monitored for at least 5 minutes until they returned to baseline values. The session duration was planned in accordance with the literature, consisting of three phases: a warm-up phase, a loading phase, and a cool-down phase, lasting a minimum of 30 minutes and a maximum of 40 minutes.
  Interventions: Other: aerobic exercise intervention

INTERVENTIONS:
Other: aerobic exercise intervention — The aerobic exercise programme was implemented over a total of 8 weeks, with two sessions per week, using a treadmill under the supervision of a specialist physiotherapist. Patients' functional capacities were determined by estimating VO2 peak using walking distance, heart rate, and blood pressure measured at 6 DYT. During the aerobic exercise programme, patients' heart rates and oxygen saturation levels were monitored using a pulse oximeter, and care was taken to ensure that the Borg Scale value perceived by patients was between 11 and 14. After the aerobic exercise programme ended, heart rate, blood pressure, and Borg Scale were monitored for at least 5 minutes until they returned to baseline values. The session duration was planned in accordance with the literature, consisting of three phases: a warm-up phase, a loading phase, and a cool-down phase, lasting a minimum of 30 minutes and a maximum of 40 minutes.
  Arms: aerobic exercise

SUMMARY:
This study is a randomised controlled trial designed to thoroughly investigate the effects of aerobic exercise on NVU biomarkers in individuals with MS. The study was conducted between February and June 2025 at the MS clinic affiliated with the Department of Neurology, Faculty of Medicine, Ondokuz Mayıs University. Participants were randomly assigned to either a control group or an exercise group. Assessments were conducted at baseline (pre-assessment) and eight weeks after the intervention (post-assessment).

DETAILED DESCRIPTION:
In multiple sclerosis (MS), impairments occur in many of the cell types involved in the functioning of the Neurovascular Unit (NVU). The study examined the relationship between aerobic exercise and biomarkers associated with NVU function in individuals with MS, including Neurofilament Light Chain (NfL), Vascular Endothelial Growth Factor (VEGF), Glial Fibrillary Acidic Protein (GFAP), and the effects of aerobic exercise on the 6-Minute Walk Test (6MWT), Timed Up and Go Test (TUG), and 9-Hole Peg Test (9HPT), which determine clinical progression.

Methods: Thirty RRMS patients with a confirmed diagnosis of MS who met the inclusion criteria were included in the study. Patients who scored 24 points or higher on the Standardised Mini Mental Test (SMMT) and had an EDSS score between 0 and 4 underwent pre-testing, which included a demographic data form, 6 DWT, TWT, and 9 DPT. Blood samples were collected for analysis of NfL, VEGF, and GFAP biomarkers. Patients were randomly assigned to either the control or exercise group, and the exercise group underwent an aerobic exercise programme for 8 weeks. After the exercise programme, all patients underwent the 6 DYT, ZKYT, and 9 DPT as a post-test, and blood samples were collected.

ELIGIBILITY:
Inclusion Criteria:

* Having a definite diagnosis of MS according to McDonald criteria,
* Being aged between 20 and 50,
* Having a Standardised Mini Mental Test (SMMT) score of ≥24,
* Having an Expanded Disability Status Scale (EDSS) score between 0 and 4.0,
* Having no other serious health problems that would prevent exercise,
* Having had no change in medication in the last 6 months.

Exclusion Criteria:

* Having experienced an MS relapse within the last 6 months,
* Having an orthopaedic or systemic problem that would prevent participation in the exercises,
* Having another known neuromuscular disorder besides MS,
* Having received immunomodulatory treatment within the last 6 months,
* Having a cardiopulmonary disorder that could prevent participation in the exercise,
* Being pregnant or breastfeeding.

Criteria for exclusion from the study:

* Failure to attend three consecutive sessions of the exercise programme
* Change in ongoing pharmacological treatment or discontinuation of pharmacological treatment
* Development of a history of MS attacks or deterioration in health status

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
clinical progression | From enrollment to the end of treatment at 8 weeks
  The primary outcome of the study is to determine clinical progression in individuals with MS. Functional mobility, walking capacity, and upper extremity functions were measured to assess clinical progression. To this end, the 6-Minute Walk Test (6MWT), 9-Hole Peg Test (9HPT), and Timed Up and Go Test (TUG) were administered. In the E group, a significant decrease was observed in dominant and non-dominant DDPT times and TWT time, while a significant increase was observed in 6WWT distance (p<0.001). No significant change was observed in these parameters in the control group (p>0.05). In the intergroup comparison, the improvements in the Exercise Group were found to be statistically significantly more pronounced than in the control group (p<0.001). These findings indicate that an eight-week aerobic exercise programme has a positive effect on clinical progression markers in individuals with MS.

SECONDARY OUTCOMES:
Neurovascular unit biomarkers | From enrollment to the end of treatment at 8 weeks
  Secondary outcomes are biomarkers reflecting NVU function. Serum NfL, serum VEGF-a, and serum GFAP were measured as NVU markers. Measurements were performed using the ELISA method with blood samples taken in the morning after all participants had fasted.
  Secondary outcome analyses revealed no significant change in NfL, VEGF-a, and GFAP levels in either within-group or between-group comparisons (p>0.05). This finding indicates that the eight-week aerobic exercise programme did not have a significant effect on NVU biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The primary reason for not sharing individual participant data (IPD) from this study is the need to ensure the highest level of data privacy and participant confidentiality. It was determined that the data could not be fully anonymized without leaving a potential risk of re-identification; therefore, IPD will not be shared. In addition, the study protocol and ethics committee approval do not include the sharing of individual-level data. However, summary-level results from the study may be shared with researchers upon reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT07325019/Prot_SAP_000.pdf